CLINICAL TRIAL: NCT02706951
Title: A Phase 3, Randomized, Double-Blind Study Comparing Upadacitinib (ABT-494) Monotherapy to Methotrexate (MTX) in Adults With Moderately to Severely Active Rheumatoid Arthritis With Inadequate Response to MTX
Brief Title: A Study Comparing Upadacitinib (ABT-494) Monotherapy to Methotrexate (MTX) Monotherapy in Adults With Rheumatoid Arthritis (RA) Who Have an Inadequate Response to MTX (SELECT-MONOTHERAPY)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-555; 2015-003376-75 (EudraCT Number)
Record Dates: First submitted 2016-02-18; First posted 2016-03-11 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Musculoskeletal Disease; Arthritis; Joint Disease; Anti-inflammatory agents; Antirheumatic agents; Upadacitinib; ABT-494
MeSH Terms: conditions — Arthritis, Rheumatoid; Musculoskeletal Diseases; Arthritis; Joint Diseases | interventions — Methotrexate; upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Upadacitinib 30 mg (Experimental): Period 1: Participants receive upadacitnib 30 mg once daily and placebo to methotrexate once weekly for 14 weeks.
  Period 2: Participants receive upadacitinib 30 mg once daily until implementation of Protocol Amendment 5 when participants begin to receive upadacitinib 15 mg once daily up to Week 260.
  Interventions: Drug: Upadacitinib; Drug: Placebo Methotrexate
- Upadacitinib 15 mg (Experimental): Period 1: Participants receive upadacitnib 15 mg once daily and placebo to methotrexate once weekly for 14 weeks.
  Period 2: Participants receive upadacitinib 15 mg once daily up to Week 260.
  Interventions: Drug: Upadacitinib; Drug: Placebo Methotrexate
- Methotrexate / Upadacitinib 30 mg (Experimental): Period 1: Participants receive methotrexate once weekly and placebo to upadacitinib once daily for 14 weeks.
  Period 2: Participants receive upadacitinib 30 mg once daily until implementation of Protocol Amendment 5 when participants begin to receive upadacitinib 15 mg once daily up to Week 260.
  Interventions: Drug: Methotrexate; Drug: Upadacitinib; Drug: Placebo Upadacitinib; Drug: Placebo Methotrexate
- Methotrexate / Upadacitinib 15 mg (Experimental): Period 1: Participants receive methotrexate once weekly and placebo to upadacitinib for 14 weeks.
  Period 2: Participants receive upadacitinib 15 mg once daily up to Week 260.
  Interventions: Drug: Methotrexate; Drug: Upadacitinib; Drug: Placebo Upadacitinib; Drug: Placebo Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Capsule; Oral
  Arms: Methotrexate / Upadacitinib 15 mg; Methotrexate / Upadacitinib 30 mg
Drug: Upadacitinib — Tablet; Oral
  Other Names: ABT-494; Rinvoq
Drug: Placebo Upadacitinib — Tablet; Oral
  Arms: Methotrexate / Upadacitinib 15 mg; Methotrexate / Upadacitinib 30 mg
Drug: Placebo Methotrexate — Capsule; Oral

SUMMARY:
The study objective of Period 1 of this study is to compare the safety and efficacy (signs and symptoms) of upadacitinib 30 mg once daily (QD) alone and upadacitinib 15 mg QD alone versus continuing MTX alone adults with moderately to severely active rheumatoid arthritis (RA) with an inadequate response to MTX.

The study objective of Period 2 is to evaluate the long term safety, tolerability, and efficacy of upadacitinib 30 mg QD and 15 mg QD in adults with RA who had completed Period 1.

DETAILED DESCRIPTION:
The study includes a 35-day screening period; a 14-week randomized, double-blind, parallel-group, controlled treatment period (Period 1); a 246-week blinded extension period (Period 2); and a 30-day follow-up visit.

Participants who met eligibility criteria were to be randomized in a 2:2:1:1 ratio to one of four treatment groups:

* Group 1: upadacitinib 30 mg QD (Period 1) → upadacitinib 30 mg QD (Period 2)
* Group 2: upadacitinib 15 mg QD (Period 1) → upadacitinib 15 mg QD (Period 2)
* Group 3: MTX (Period 1) → upadacitinib 30 mg QD (Period 2)
* Group 4: MTX (Period 1) → upadacitinib 15 mg QD (Period 2)

Starting with implementation of Protocol Amendment 5, all participants in the extension period will receive open-label upadacitinib 15 mg QD, including those currently on upadacitinib 30 mg QD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA for >= 3 months.
* Subjects must have been on oral or parenteral MTX therapy >= 3 months and on a stable dose for >= 4 weeks prior to first dose of study drug.
* Must have discontinued all conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs) (other than MTX) >= 4 weeks prior to first dose of study drug.
* Meets the following minimum disease activity criteria: >= 6 swollen joints (based on 66 joint counts) and >= 6 tender joints (based on 68 joint counts) at Screening and Baseline Visits.

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor (including but not limited to tofacitinib, baricitinib, and filgotinib).
* Prior exposure to any biological disease-modifying anti-rheumatic drugs (bDMARDs).
* Current diagnosis of inflammatory joint disease other than RA. Current diagnosis of secondary Sjogren's Syndrome is permitted.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2022-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (153):
- United States (52):
  - Rheum Assoc of North Alabama /ID# 146009, Huntsville, Alabama
  - Alabama Medical Group, PC /ID# 153941, Mobile, Alabama
  - ArthroCare Arthritis Care & Re /ID# 143751, Gilbert, Arizona
  - Elite Clinical Studies, LLC /ID# 143760, Phoenix, Arizona
  - University of Arizona Cancer Center - North Campus /ID# 147175, Tucson, Arizona
  - NEA Baptist Womens Clinic /ID# 148904, Jonesboro, Arkansas
  - C.V. Mehta MD, Med Corporation /ID# 143762, Hemet, California
  - Arthritis Assoc & Osteo Ctr /ID# 147176, Colorado Springs, Colorado
  - Ctr Rheum, Immuno, Arthritis /ID# 143766, Fort Lauderdale, Florida
  - South Florida Research Ph I-IV /ID# 151983, Miami Springs, Florida
  - Advent Clinical Research /ID# 143767, Pinellas Park, Florida
  - Sarasota Arthritis Center /ID# 146011, Sarasota, Florida
  - W. Broward Rheum Assoc Inc. /ID# 146010, Tamarac, Florida
  - Clinical Research West FL /ID# 148726, Tampa, Florida
  - SW FL Clin Res Ctr, Tampa, FL /ID# 143763, Tampa, Florida
  - University of South Florida /ID# 146004, Tampa, Florida
  - BayCare Medical Group, Inc. /ID# 151985, Tampa, Florida
  - BayCare Medical Group, Inc. /ID# 163595, Tampa, Florida
  - Jefrey D. Lieberman, MD, P.C. /ID# 151816, Decatur, Georgia
  - Great Lakes Clinical Trials /ID# 150935, Chicago, Illinois
  - PRN Professional Research Network of Kansas, LLC /ID# 143761, Wichita, Kansas
  - Ochsner Clinic Foundation /ID# 153573, Baton Rouge, Louisiana
  - The Arthritis & Diabetes Clinic, Inc. /ID# 160809, Monroe, Louisiana
  - Vanguard Medical Research, LLC /ID# 153124, Shreveport, Louisiana
  - Mansfield Health Center /ID# 161627, Mansfield, Massachusetts
  - Quality Clinical Research Inc. /ID# 156415, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center /ID# 146008, Lebanon, New Hampshire
  - Albuquerque Clinical Trials, Inc /ID# 147618, Albuquerque, New Mexico
  - Arthritis and Osteo Assoc /ID# 147177, Las Cruces, New Mexico
  - Coastal Carolina Health Care /ID# 149275, New Bern, North Carolina
  - STAT Research, Inc. /ID# 143770, Vandalia, Ohio
  - Health Research Oklahoma /ID# 159550, Oklahoma City, Oklahoma
  - Healthcare Research Consultant /ID# 147632, Tulsa, Oklahoma
  - Innovative Clinical Research /ID# 143757, Greenville, South Carolina
  - Nashville Arthritis and Rheumatology /ID# 162641, Nashville, Tennessee
  - Tekton Research, Inc. /ID# 159554, Austin, Texas
  - Diagnostic Group Integrated He /ID# 148725, Beaumont, Texas
  - Trinity Universal Res Assoc /ID# 150138, Carrollton, Texas
  - Arth and Osteo Clin Brazo Valley /ID# 160810, College Station, Texas
  - Adriana Pop-Moody MD Clinic PA /ID# 147627, Corpus Christi, Texas
  - Accurate Clinical Management /ID# 143768, Houston, Texas
  - Accurate Clinical Research /ID# 143769, Houston, Texas
  - Pioneer Research Solutions, Inc. /ID# 143765, Houston, Texas
  - P&I Clinical Research /ID# 151358, Lufkin, Texas
  - SW Rheumatology Res. LLC /ID# 147620, Mesquite, Texas
  - Sun Research Institute /ID# 159553, San Antonio, Texas
  - Arthritis Clinic of Central TX /ID# 149266, San Marcos, Texas
  - Adv Rheumatology of Houston /ID# 162609, The Woodlands, Texas
  - DM Clinical Research /ID# 151359, Tomball, Texas
  - Arthritis & Osteoporosis Clinic /ID# 143752, Waco, Texas
  - Ctr for Arth and Rheum Disease /ID# 143759, Chesapeake, Virginia
  - Aurora Rheumatology and Immunotherapy Center /ID# 160811, Franklin, Wisconsin
- Argentina (6):
  - Mautalen Salud e Investigacion /ID# 145980, Buenos Aires
  - Ctr Privado Med Familiar /ID# 149183, Buenos Aires
  - Consultorio Reumatologic Pampa /ID# 145979, Buenos Aires
  - Centro de Educación Médica e Investigaciones Clínicas "Norberto Quimo" - CEMIC /ID# 149176, Buenos Aires
  - Cordis S.A. /Id# 152621, Salta
  - Centro de Enfermedades /ID# 153543, Santa Fe
- Royal Prince Alfred Hospital /ID# 146028, Camperdown, New South Wales, Australia
- Rheuma-Zentrum Wien-Oberlaa /ID# 144728, Vienna, Austria
- Belgium (2):
  - Algemeen Stedelijk Ziekenhuis /ID# 148720, Aalst, Oost-Vlaanderen
  - ReumaClinic Genk /ID# 146030, Genk
- Bulgaria (2):
  - Diag Consult Ctr 17 Sofia EOOD /ID# 144730, Sofia
  - UMHAT Sv. Ivan Rilski /ID# 147351, Sofia
- Chile (3):
  - Reg. Clinical Hosptial Concepcion /ID# 151267, Concepción
  - Quantum Research LTDA. /ID# 145984, Puerto Varas
  - Quantum Research Stgo. /ID# 145983, Santiago
- Czechia (5):
  - CTCenter MaVe, s.r.o. /ID# 144823, Olomouc, Olomoucký kraj
  - Nuselská poliklinika, Revmatologie /ID# 145986, Prague, Praha 4
  - Thomayerova nemocnice /ID# 144736, Prague, Praha 4
  - RHEUMA s.r.o. /ID# 144737, Břeclav
  - Medical Plus, s.r.o. /ID# 144821, Uherské Hradište
- Estonia (2):
  - MediTrials /ID# 159745, Tartu, Tartu
  - North Estonian Medical Centre /ID# 145455, Tallinn
- General Hospital of Athens "Ippokratio" /ID# 144739, Athens, Greece
- Hungary (4):
  - Vital Medical Center Orvosi es /ID# 144740, Veszprém, Veszprém megye
  - Magyar Honvedseg Egeszsegugyi Kozpont /ID# 144743, Budapest
  - Pest Megyei Flor Ferenc Korhaz /ID# 144742, Kistarcsa
  - Fejer Megyei Szent Gyorgy Korh /ID# 144741, Székesfehérvár
- Israel (4):
  - Barzilai Medical Center /ID# 144744, Ashkelon
  - Bnai Zion Medical Center /ID# 144745, Haifa
  - The Lady Davis Carmel MC /ID# 147174, Haifa
  - Sheba Medical Center /ID# 144824, Ramat Gan
- Italy (2):
  - Universita di Catanzaro Magna Graecia /ID# 144747, Catanzaro, Calabria
  - A.O.U.I. di Verona Policlinico /ID# 144746, Verona
- Japan (21):
  - Kondo Clinic for Rheum & Ortho /ID# 148268, Fukuoka, Fukuoka
  - NHO Kyushu Medical Center /ID# 148279, Fukuoka, Fukuoka
  - NHO Kyushu Medical Center /ID# 148280, Fukuoka, Fukuoka
  - Aso Iizuka Hospital /ID# 148272, Iizuka-shi, Fukuoka
  - Inoue Hospital /ID# 148069, Takasaki, Gunma
  - Bay Side Misato Medical Center /ID# 148281, Kochi, Kochi
  - Center for Arthritis and Clinical Rheumatology Matsubara Clinic /ID# 148269, Kumamoto, Kumamoto
  - Kumamoto Shinto General Hospital /ID# 148286, Kumamoto, Kumamoto
  - Nagasaki University Hospital /ID# 149859, Nagasaki, Nagasaki
  - Sasebo Chuo Hospital /ID# 148275, Sasebo, Nagasaki
  - Osaka Red Cross Hospital /ID# 148267, Osaka, Osaka
  - Seirei Hamamatsu General Hosp /ID# 148270, Hamamatsu
  - Ohira Orthopaedic Hospital /ID# 157944, Hyūga
  - Shirahama Hamayu Hospital /ID# 148277, Nishimura
  - Sanuki Municipal Hospital /ID# 158080, Sanuki
  - Hokkaido University Hospital /ID# 148285, Sapporo
  - Hokkaido Medical Center for Rheumatic Diseases /ID# 148274, Sapporo
  - Miyasato Clinic /ID# 148271, Shūnan
  - Takaoka Rheumatic Orthopedic Clinic /ID# 148068, Takaoka
  - Matsuta Clinic /ID# 148278, Tokyo
  - National Hospital Organization Shimoshizu National Hospital /ID# 148273, Yotsukaidō
- Mexico (2):
  - Desarrollos Biomedicos y Biotc /ID# 147379, Monterrey, Nuevo León
  - Cryptex Investigación Clínica S.A de C.V /ID# 147095, Mexico City
- Poland (7):
  - Medyczne Centrum Hetmanska /ID# 144751, Poznan, Greater Poland Voivodeship
  - WroMedica I. Bielicka, A. Strzalkowska s.c. /ID# 157622, Wroclaw, Lower Silesian Voivodeship
  - REUMED Sp.z o.o. Filia nr 1 /ID# 144752, Lublin, Lublin Voivodeship
  - Centralny Szpital Kliniczny MSWiA w Warszawie /ID# 149521, Warsaw, Masovian Voivodeship
  - Osteo-Medic spolka cywilna /ID# 144753, Bialystok, Podlaskie Voivodeship
  - Centrum Badań Klinicznych Pi-House /ID# 149520, Gdansk, Pomeranian Voivodeship
  - NZOZ Centrum Reumatologiczne /ID# 144749, Elblag, Warmian-Masurian Voivodeship
- Portugal (4):
  - Instituto Portugues De Reumatologia /ID# 149281, Lisbon, Lisbon District
  - Centro Hospitalar De Vila Nova /ID# 146036, Vila Nova de Gaia, Porto District
  - Centro Hospitalar Lisboa Norte, EPE /ID# 146035, Lisbon
  - Centro Hospitalar Baixo Vouga /ID# 152916, Porto
- Puerto Rico (2):
  - Dr. Ramon L. Ortega-Colon, MD /ID# 145989, Carolina
  - Ponce School of Medicine /ID# 145990, Ponce
- Spitalul Municipal Ploiesti /ID# 144756, Ploieşti, Romania
- Russia (12):
  - Clinical Hospital No.1 n.a. N.I.Pirogov /ID# 147255, Moscow, Moscow
  - LLC Medical Center /ID# 144758, Novosibirsk, Novosibirsk Oblast
  - Perm Clinical Center of FMBA /ID# 145993, Perm, Permskiy Kray
  - Tver Regional Clinical Hosp. /ID# 147254, Tver', Tver Oblast
  - Сity Clinical Hospital 4 /ID# 145994, Ivanovo
  - City Clinical Hospital Botkina /ID# 145995, Moscow
  - City Clinical Hospital #5 /ID# 149832, Nizhny Novgorod
  - Orenburg State Medical Academy /ID# 145992, Orenburg
  - Republican Clin Hos n.a. Baran /ID# 147251, Petrozavodsk
  - Samara Regional Clinical Hosp /ID# 150934, Samara
  - Reg Clin Hosp n.a. Kuvatova G. /ID# 144757, Ufa
  - Yaroslavi State Medical Univer /ID# 147253, Yaroslavl
- Serbia (4):
  - Institute for Rheumatology /ID# 144759, Belgrade, Beograd
  - Institute for Rheumatology /ID# 144761, Belgrade, Beograd
  - Institute for Rheumatology /ID# 144762, Belgrade, Beograd
  - Special Hospital for Rheuma /ID# 144760, Novi Sad, Vojvodina
- South Africa (4):
  - Wits Clinical Research Site /ID# 149835, Johannesburg, Gauteng
  - University of Pretoria /ID# 148740, Pretoria, Gauteng
  - Synexus Helderberg Clinical Tr /ID# 148724, Cape Town, Western Cape
  - Tiervlei Trial Centre /ID# 153086, Cape Town, Western Cape
- Spain (5):
  - Hospital Plató /ID# 145999, Barcelona
  - Hospital Univ Germans Trias I /ID# 146037, Barcelona
  - Hospital Infanta Luisa /ID# 144771, Seville
  - Hospital Universitario de Valm /ID# 144770, Seville
  - Hospital Universitario La Fe /ID# 158013, Valencia
- Uludağ Üniversitesi Atatürk Rehabilitasyon Uygulama ve Araştırma Merkezi /ID# 144772, Osmangazi, Bursa, Turkey (Türkiye)
- Ukraine (5):
  - Lviv Regional Clinical Hospita /ID# 154448, Lviv, Lviv Oblast
  - Vinnytsia Regional Clinical Hospital n.a. M.I.Pyrogov /ID# 146002, Vinnytsia, Vinnytsia Oblast
  - Regional Clinical Hospital /ID# 152007, Ivano-Frankivsk
  - NSC-Strazhesko Ist Cardiology /ID# 152004, Kiev
  - Zaporizhzhia Regional Clinical /ID# 146000, Zaporizhia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Background] Smolen JS, Pangan AL, Emery P, Rigby W, Tanaka Y, Vargas JI, Zhang Y, Damjanov N, Friedman A, Othman AA, Camp HS, Cohen S. Upadacitinib as monotherapy in patients with active rheumatoid arthritis and inadequate response to methotrexate (SELECT-MONOTHERAPY): a randomised, placebo-controlled, double-blind phase 3 study. Lancet. 2019 Jun 8;393(10188):2303-2311. doi: 10.1016/S0140-6736(19)30419-2. Epub 2019 May 23. PMID 31130260
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Smolen JS, Emery P, Rigby W, Tanaka Y, Vargas JI, Jain M, Kato K, Carter KM, Khan N, Phillips C, Meerwein S, Cohen SB. Upadacitinib as monotherapy in patients with rheumatoid arthritis and prior inadequate response to methotrexate: results at 260 weeks from the SELECT-MONOTHERAPY randomised study. RMD Open. 2025 May 11;11(2):e005051. doi: 10.1136/rmdopen-2024-005051. PMID 40350200
- [Derived] Rubbert-Roth A, Kakehasi AM, Takeuchi T, Schmalzing M, Palac H, Coombs D, Liu J, Anyanwu SI, Lippe R, Curtis JR. Malignancy in the Upadacitinib Clinical Trials for Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis, and Non-radiographic Axial Spondyloarthritis. Rheumatol Ther. 2024 Feb;11(1):97-112. doi: 10.1007/s40744-023-00621-6. Epub 2023 Nov 20. PMID 37982966
- [Derived] Charles-Schoeman C, Choy E, McInnes IB, Mysler E, Nash P, Yamaoka K, Lippe R, Khan N, Shmagel AK, Palac H, Suboticki J, Curtis JR. MACE and VTE across upadacitinib clinical trial programmes in rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis. RMD Open. 2023 Nov;9(4):e003392. doi: 10.1136/rmdopen-2023-003392. PMID 37945286
- [Derived] Fleischmann R, Curtis JR, Charles-Schoeman C, Mysler E, Yamaoka K, Richez C, Palac H, Dilley D, Liu J, Strengholt S, Burmester G. Safety profile of upadacitinib in patients at risk of cardiovascular disease: integrated post hoc analysis of the SELECT phase III rheumatoid arthritis clinical programme. Ann Rheum Dis. 2023 Sep;82(9):1130-1141. doi: 10.1136/ard-2023-223916. Epub 2023 Jun 12. PMID 37308218
- [Derived] Conaghan PG, Pavelka K, Hsieh SC, Bonnington TL, Kent TC, Marchbank K, Edwards CJ. Evaluating the efficacy of upadacitinib in patients with moderate rheumatoid arthritis: a post-hoc analysis of the SELECT phase 3 trials. Rheumatol Adv Pract. 2023 Feb 8;7(1):rkad017. doi: 10.1093/rap/rkad017. eCollection 2023. PMID 36794283
- [Derived] Burmester GR, Cohen SB, Winthrop KL, Nash P, Irvine AD, Deodhar A, Mysler E, Tanaka Y, Liu J, Lacerda AP, Palac H, Shaw T, Mease PJ, Guttman-Yassky E. Safety profile of upadacitinib over 15 000 patient-years across rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and atopic dermatitis. RMD Open. 2023 Feb;9(1):e002735. doi: 10.1136/rmdopen-2022-002735. PMID 36754548
- [Derived] Kakehasi AM, Radominski SC, Baravalle MD, Palazuelos FCI, Garcia-Garcia C, Arruda MS, Curi M, Liu J, Qiao M, Velez-Sanchez P, Vargas JI. Safety of upadacitinib in Latin American patients with rheumatoid arthritis: an integrated safety analysis of the SELECT phase 3 clinical program. Clin Rheumatol. 2023 May;42(5):1249-1258. doi: 10.1007/s10067-023-06513-y. Epub 2023 Jan 30. PMID 36715850
- [Derived] Bergman M, Buch MH, Tanaka Y, Citera G, Bahlas S, Wong E, Song Y, Zueger P, Ali M, Strand V. Routine Assessment of Patient Index Data 3 (RAPID3) in Patients with Rheumatoid Arthritis Treated with Long-Term Upadacitinib Therapy in Five Randomized Controlled Trials. Rheumatol Ther. 2022 Dec;9(6):1517-1529. doi: 10.1007/s40744-022-00483-4. Epub 2022 Sep 20. PMID 36125701
- [Derived] Bergman M, Tundia N, Yang M, Orvis E, Clewell J, Bensimon A. Economic Benefit from Improvements in Quality of Life with Upadacitinib: Comparisons with Tofacitinib and Methotrexate in Patients with Rheumatoid Arthritis. Adv Ther. 2021 Dec;38(12):5649-5661. doi: 10.1007/s12325-021-01930-4. Epub 2021 Oct 12. PMID 34636000
- [Derived] Yamaoka K, Tanaka Y, Kameda H, Khan N, Sasaki N, Harigai M, Song Y, Zhang Y, Takeuchi T. The Safety Profile of Upadacitinib in Patients with Rheumatoid Arthritis in Japan. Drug Saf. 2021 Jun;44(6):711-722. doi: 10.1007/s40264-021-01067-x. Epub 2021 May 27. PMID 34041702
- [Derived] Strand V, Tundia N, Wells A, Buch MH, Radominski SC, Camp HS, Friedman A, Suboticki JL, Dunlap K, Goldschmidt D, Bergman M. Upadacitinib monotherapy improves patient-reported outcomes in rheumatoid arthritis: results from SELECT-EARLY and SELECT-MONOTHERAPY. Rheumatology (Oxford). 2021 Jul 1;60(7):3209-3221. doi: 10.1093/rheumatology/keaa770. PMID 33313898
- [Derived] Cohen SB, van Vollenhoven RF, Winthrop KL, Zerbini CAF, Tanaka Y, Bessette L, Zhang Y, Khan N, Hendrickson B, Enejosa JV, Burmester GR. Safety profile of upadacitinib in rheumatoid arthritis: integrated analysis from the SELECT phase III clinical programme. Ann Rheum Dis. 2021 Mar;80(3):304-311. doi: 10.1136/annrheumdis-2020-218510. Epub 2020 Oct 28. PMID 33115760
- [Derived] Nader A, Mohamed MF, Winzenborg I, Doelger E, Noertersheuser P, Pangan AL, Othman AA. Exposure-Response Analyses of Upadacitinib Efficacy and Safety in Phase II and III Studies to Support Benefit-Risk Assessment in Rheumatoid Arthritis. Clin Pharmacol Ther. 2020 Apr;107(4):994-1003. doi: 10.1002/cpt.1671. Epub 2019 Nov 30. PMID 31610021
- See also: Related Info. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 648 participants with rheumatoid arthritis (RA) on a stable dose of methotrexate (MTX) were randomized at 138 study sites located in 24 countries.
Pre-assignment Details: Participants were randomized in a 2:2:1:1 ratio to 1 of 4 groups:
  * Upadacitinib 30 mg (Periods 1 and 2)
  * Upadacitinib 15 mg (Periods 1 and 2)
  * MTX (Period 1) → upadacitinib 30 mg (Period 2)
  * MTX (Period 1) → upadacitinib 15 mg (Period 2)
  Randomization was stratified by geographic region. The MTX groups were pooled for Week 14 analyses.
  Starting with Amend. 5 & during Period 2, all participants received open-label upadacitinib 15 mg, including participants receiving upadacitinib 30 mg
Groups:
- Period 1: Methotrexate: Participants randomized to receive up to 25 mg methotrexate once a week and placebo to upadacitinib once daily (QD) for 14 weeks in Period 1.
- Period 1: Upadacitinib 15 mg: Participants randomized to receive upadacitinib 15 mg once daily and placebo to methotrexate once a week for 14 weeks in Period 1.
- Period 1: Upadacitinib 30 mg: Participants randomized to receive upadacitinib 30 mg once daily and placebo to methotrexate once a week for 14 weeks in Period 1.
- Period 2: Upadacitinib 15 mg: Continuing Period 1 participants that were randomized into the upadacitinib 15 mg once daily arm combined with Period 1 Methotrexate (MTX) participants that were randomized to receive upadacitinib 15 mg once daily in Period 2
- Period 2: Upadacitinib 30 mg: Continuing Period 1 participants that were randomized into the upadacitinib 30 mg once daily arm combined with Period 1 Methotrexate (MTX) participants that were randomized to receive upadacitinib 30 mg once daily in Period 2
Period: Period 1
Arm/Group | Period 1: Methotrexate | Period 1: Upadacitinib 15 mg | Period 1: Upadacitinib 30 mg | Period 2: Upadacitinib 15 mg | Period 2: Upadacitinib 30 mg
Started | 216 | 217 | 215 | 0 | 0
Completed (Completed Period 1 (Week 14) study participation) | 203 | 201 | 205 | 0 | 0
Not Completed | 13 | 16 | 10 | 0 | 0
Not completed — Adverse Event | 1 | 5 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 6 | 6 | 0 | 0
Not completed — Lost to Follow-up | 0 | 4 | 1 | 0 | 0
Not completed — Other | 2 | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Period 1: Methotrexate | Period 1: Upadacitinib 15 mg | Period 1: Upadacitinib 30 mg | Period 2: Upadacitinib 15 mg | Period 2: Upadacitinib 30 mg
Started | 0 | 0 | 0 | 302 | 300
Completed | 0 | 0 | 0 | 184 | 180
Not Completed | 0 | 0 | 0 | 118 | 120
Not completed — Adverse Event | 0 | 0 | 0 | 25 | 34
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 38 | 44
Not completed — Lost to Follow-up | 0 | 0 | 0 | 17 | 9
Not completed — COVID-19 Related | 0 | 0 | 0 | 1 | 2
Not completed — Other | 0 | 0 | 0 | 37 | 31

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug.
Groups:
- Methotrexate: Participants randomized to receive up to 25 mg methotrexate once a week and placebo to upadacitinib once daily for 14 weeks in Period 1.
- Upadacitinib 15 mg: Participants randomized to receive upadacitinib 15 mg once daily and placebo to methotrexate once a week for 14 weeks in Period 1.
- Upadacitinib 30 mg: Participants randomized to receive upadacitinib 30 mg once daily and placebo to methotrexate once a week for 14 weeks in Period 1.
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg | Total
Number analyzed (Participants) | 216 | 217 | 215 | 648
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (11.12) | 54.5 (12.20) | 53.1 (12.72) | 54.3 (12.05)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 23 | 28 | 31 | 82
  40 - 64 years | 148 | 147 | 141 | 436
  ≥ 65 years | 45 | 42 | 43 | 130
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 174 | 170 | 523
  Male | 37 | 43 | 45 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 52 | 54 | 156
  Not Hispanic or Latino | 166 | 165 | 161 | 492
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 176 | 173 | 180 | 529
  Black or African American | 11 | 15 | 9 | 35
  American Indian/Alaska Native | 3 | 4 | 3 | 10
  Asian | 24 | 24 | 21 | 69
  Multiple | 2 | 1 | 2 | 5
Geographic Region [Count of Participants; unit: Participants] — Other includes South Africa, Turkey, and Israel.
  Participants
    North America | 64 | 64 | 64 | 192
    South/Central America | 31 | 30 | 30 | 91
    Western Europe | 8 | 8 | 8 | 24
    Eastern Europe | 79 | 80 | 80 | 239
    Asia - Japan | 22 | 22 | 21 | 65
    Other | 12 | 13 | 12 | 37
Duration of RA Diagnosis [Mean (Standard Deviation); unit: years] | 5.8 (6.63) | 7.5 (8.88) | 6.5 (6.98) | 6.6 (7.58)
Tender Joint Count [Mean (Standard Deviation); unit: joints] — A total of 68 joints were assessed for the presence or absence of tenderness.
  joints | 25.2 (15.99) | 24.5 (15.10) | 24.8 (15.19) | 24.8 (15.41)
Swollen Joint Count [Mean (Standard Deviation); unit: joints] — A total of 66 joints were assessed for the presence or absence of swelling.
  joints | 16.9 (11.52) | 16.4 (10.94) | 16.9 (10.23) | 16.7 (10.90)
Patient's Assessment of Pain [Mean (Standard Deviation); unit: mm] — Participants were asked to indicate the severity of their arthritis pain within the previous week on a visual analog scale (VAS) from 0 to 100 mm. A score of 0 mm indicates "no pain" and a score of 100 mm indicates "worst possible pain." Population: Participants with available data
  mm
    number analyzed (Participants) | 216 | 216 | 215 | 647
    (all) | 62.5 (21.26) | 62.3 (22.53) | 61.9 (22.12) | 62.3 (21.94)
Patient's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — The participant was asked to rate their current RA disease activity over the past 24 hours on a 100 mm VAS, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity. Population: Participants with available data
  mm
    number analyzed (Participants) | 216 | 216 | 215 | 647
    (all) | 59.6 (21.78) | 62.2 (22.29) | 59.4 (22.79) | 60.4 (22.29)
Physician's Global Assessment of Disease Activity [Mean (Standard Deviation); unit: mm] — The physician rated the participant's current global RA disease activity (independently from the participant's assessment) on a VAS scale from 0 to 100 mm, where 0 mm indicates very low disease activity and 100 mm indicates very high disease activity. Population: Participants with available data
  mm
    number analyzed (Participants) | 200 | 209 | 202 | 611
    (all) | 62.1 (17.47) | 65.7 (18.49) | 62.6 (17.81) | 63.5 (17.98)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 216 | 216 | 215 | 647
    (all) | 1.5 (0.66) | 1.5 (0.66) | 1.5 (0.65) | 1.5 (0.66)
High-sensitivity C-reactive Protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] | 14.5 (17.33) | 14.0 (16.49) | 16.3 (20.77) | 14.9 (18.28)
Disease Activity Score 28 Based on CRP (DAS28[CRP]) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L).
  Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A DAS28 score > 5.1 indicates high disease activity, a DAS28 score ≤ 3.2 indicates low disease activity, and a DAS28 score < 2.6 indicates clinical remission. Population: Participants with available data
  units on a scale
    number analyzed (Participants) | 216 | 216 | 215 | 647
    (all) | 5.6 (1.04) | 5.6 (0.92) | 5.6 (1.06) | 5.6 (1.01)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 14
Description: The primary endpoint for United States (US)/Food and Drug Administration (FDA) regulatory purposes was ACR 20% response (ACR20) at Week 14. Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR20 response criteria:
  1. ≥ 20% improvement in 68-tender joint count;
  2. ≥ 20% improvement in 66-swollen joint count; and
  3. ≥ 20% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and week 14
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 14 or for whom ACR data were missing at Week 14 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 216 | 217 | 215
percentage of participants | 41.2 [34.6 to 47.8] | 67.7 [61.5 to 74.0] | 71.2 [65.1 to 77.2]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — The overall type I error prevalence of the primary and ranked key secondary endpoints for the two doses of upadacitinib were strongly controlled by means of a graphic multiple testing procedure; p < 0.001, Cochran-Mantel-Haenszel — The adjusted p-value under multiplicity control is reported, with significance achieved if the adjusted p-value is less than 0.05; Cochran-Mantel-Haenszel test adjusted for stratification factor geographic region; Response Rate Difference = 26.5, 95% CI 2-sided [17.5 to 35.6] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel test adjusted for stratification factor geographic region; Response Rate Difference = 30.0, 95% CI 2-sided [21.0 to 38.9] — Response Rate Difference = Upadacitinib - Methotrexate

2. Primary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on DAS28(CRP) at Week 14
Description: The primary endpoint for European Union (EU)/European Medicines Agency (EMA) regulatory purposes was low disease activity, based on a Disease Activity Score 28 (DAS28)-CRP score of ≤ 3.2 at Week 14.
  The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
  A DAS28 score less than or equal to 3.2 indicates low disease activity.
Time Frame: Week 14
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 14 or for whom DAS28 data were missing at Week 14 were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 216 | 217 | 215
percentage of participants | 19.4 [14.2 to 24.7] | 44.7 [38.1 to 51.3] | 53.0 [46.4 to 59.7]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel test adjusted for stratification factor geographic region; Response Rate Difference = 25.3, 95% CI 2-sided [16.8 to 33.7] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel test adjusted for stratification factor geographic region; Response Rate Difference = 33.6, 95% CI 2-sided [25.1 to 42.1] — Response Rate Difference = Upadacitinib - Methotrexate

3. Secondary Outcome: Change From Baseline in in Disease Activity Score 28 (CRP) at Week 14
Description: The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change from baseline in DAS28 (CRP) indicates improvement in disease activity.
Time Frame: Baseline to week 14
Population: Full analysis set participants with available data at baseline; multiple imputation was used for missing post-baseline data.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 215 | 215 | 213
scores on a scale | -1.20 [-1.39 to -1.01] | -2.29 [-2.48 to -2.10] | -2.61 [-2.80 to -2.41]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Analysis of covariance (ANCOVA) model with treatment as the fixed factor, and baseline value and geographic region as the covariates; Least Squares (LS) Mean Difference = -1.08, 95% CI 2-sided [-1.32 to -0.85] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model with treatment as the fixed factor, and baseline value and the stratification factor geographic region as the covariates; LS Mean Difference = -1.40, 95% CI 2-sided [-1.64 to -1.17] — Difference = Upadacitinib - Methotrexate

4. Secondary Outcome: Change From Baseline in Heath Assessment Questionnaire and Disability Index (HAQ-DI) at Week 14
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline to week 14
Population: Full analysis set participants with available data at baseline; multiple imputation was used for missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 216 | 216 | 215
scores on a scale | -0.32 [-0.41 to -0.23] | -0.65 [-0.73 to -0.56] | -0.73 [-0.82 to -0.64]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = -0.33, 95% CI 2-sided [-0.43 to -0.22] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 2]; LS Mean Difference = -0.41, 95% CI 2-sided [-0.51 to -0.30] — Difference = Upadacitinib - Methotrexate

5. Secondary Outcome: Change From Baseline in Short-Form 36 (SF-36) Physical Component Score (PCS) at Week 14
Description: The Short Form 36-Item Health Survey (SF-36) Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component score is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The PCS was calculated using norm-based scoring so that 50 is the average score and the standard deviation equals 10. Higher scores are associated with better functioning/quality of life; a positive change from baseline score indicates an improvement.
Time Frame: Baseline to week 14
Population: Full analysis set participants with available data; a mixed effect model repeat measurement (MMRM) analysis with data from observed cases to Week 14 was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 195 | 200 | 201
scores on a scale | 4.32 [3.19 to 5.44] | 8.28 [7.17 to 9.40] | 10.19 [9.07 to 11.30]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; MMRM model with fixed effects of treatment, visit, treatment-by-visit interaction, and geographic region, and the baseline value as covariate; LS Mean Difference = 3.97, 95% CI 2-sided [2.52 to 5.42] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = 5.87, 95% CI 2-sided [4.42 to 7.32] — Difference = Upadacitinib - Methotrexate

6. Secondary Outcome: Percentage of Participants Achieving Clinical Remission (CR) Based on DAS28(CRP) at Week 14
Description: The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity.
  A DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 216 | 217 | 215
percentage of participants | 8.3 [4.6 to 12.0] | 28.1 [22.1 to 34.1] | 40.5 [33.9 to 47.0]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel test adjusted for stratification factor geographic region; Response Rate Difference = 19.8, 95% CI 2-sided [12.8 to 26.8] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Cochran-Mantel-Haenszel test adjusted for stratification factor geographic region; Response Rate Difference = 32.1, 95% CI 2-sided [24.6 to 39.7] — Response Rate Difference = Upadacitinib - Methotrexate

7. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Week 14
Description: Participants were asked to indicate the time it took for them to get as limber as possible after awakening with morning stiffness over the past 7 days. A negative change from Baseline indicates improvement.
Time Frame: Baseline to week 14
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 196 | 199 | 202
minutes | -53.03 [-72.18 to -33.88] | -94.56 [-113.57 to -75.54] | -102.34 [-121.24 to -83.45]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = -41.53, 95% CI 2-sided [-66.56 to -16.50] — Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Effect Model Repeat Measurement — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 5, analysis 1]; LS Mean Difference = -49.31, 95% CI 2-sided [-74.23 to -24.40] — Difference = Upadacitinib - Methotrexate

8. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 14
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and week 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 216 | 217 | 215
percentage of participants | 15.3 [10.5 to 20.1] | 41.9 [35.4 to 48.5] | 52.1 [45.4 to 58.8]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; the nominal p-value is reported; Cochran-Mantel-Haenszel test adjusted for stratification factor geographic region; Response Rate Difference = 26.7, 95% CI 2-sided [18.5 to 34.8] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; the nominal p-value is reported; Cochran-Mantel-Haenszel test adjusted for stratification factor geographic region; Response Rate Difference = 36.8, 95% CI 2-sided [28.6 to 45.0] — Response Rate Difference = Upadacitinib - Methotrexate

9. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 70% (ACR70) Response at Week 14
Description: Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 70% improvement in 68-tender joint count;
  2. ≥ 70% improvement in 66-swollen joint count; and
  3. ≥ 70% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and week 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methotrexate | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 216 | 217 | 215
percentage of participants | 2.8 [0.6 to 5.0] | 22.6 [17.0 to 28.1] | 33.0 [26.7 to 39.3]
Statistical Analysis 1: Comparison: Methotrexate vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; the nominal p-value is reported; Cochran-Mantel-Haenszel test adjusted for stratification factor geographic region; Response Rate Difference = 19.8, 95% CI 2-sided [13.8 to 25.8] — Response Rate Difference = Upadacitinib - Methotrexate
Statistical Analysis 2: Comparison: Methotrexate vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — This comparison was not part of the pre-specified multiplicity testing sequence; the nominal p-value is reported; Cochran-Mantel-Haenszel test adjusted for stratification factor geographic region; Response Rate Difference = 30.2, 95% CI 2-sided [23.6 to 36.9] — Response Rate Difference = Upadacitinib - Methotrexate

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Adverse Event collection in Period 2 combined the Periods 1+2 Upadacitinib 15 mg Arm which includes 101 participants who were re-randomized from the Period 1 Methotrexate Arm in addition to the 217 participants who started in the Period 1 Upadacitinib 15 mg Arm. The Upadacitinib 30 mg Arm includes 96 participants who were re-randomized from the Period 1 Methotrexate Arm in addition to the 215 participants who started in the Period 1 Upadacitinib 30 mg Arm
Groups:
- Period 1: Methotrexate: Participants randomized to receive up to 25 mg methotrexate once a week and placebo to upadacitinib once daily for 14 weeks in Period 1.
- Periods 1+2: Upadacitinib 15 mg: Participants randomized to receive upadacitinib 15 mg once daily
- Periods 1+ 2: Upadacitinib 30 mg: Participants randomized to receive upadacitinib 30 mg once daily
- Period 2: Upadacitinib 15 mg Switched From Upadacitinib 30 mg: Starting with Amendment 5, all participants will receive open-label upadacitinib 15 mg once daily, including those currently on upadacitinib 30 mg once daily
Arm/Group | Period 1: Methotrexate | Period 1: Upadacitinib 15 mg | Period 1: Upadacitinib 30 mg | Periods 1+2: Upadacitinib 15 mg | Periods 1+ 2: Upadacitinib 30 mg | Period 2: Upadacitinib 15 mg Switched From Upadacitinib 30 mg
All-Cause Mortality (participants affected / at risk) | 0/216 | 0/217 | 0/215 | 7/318 | 5/311 | 4/205
Serious Adverse Events (participants affected / at risk) | 7/216 | 11/217 | 6/215 | 95/318 | 75/311 | 22/205
Other Adverse Events (participants affected / at risk) | 49/216 | 43/217 | 51/215 | 219/318 | 211/311 | 82/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Methotrexate (N=216) | Period 1: Upadacitinib 15 mg (N=217) | Period 1: Upadacitinib 30 mg (N=215) | Periods 1+2: Upadacitinib 15 mg (N=318) | Periods 1+ 2: Upadacitinib 30 mg (N=311) | Period 2: Upadacitinib 15 mg Switched From Upadacitinib 30 mg (N=205)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone marrow oedema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mixed deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bartholin's abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 4 (4) | 7 (7)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 12 (12) | 4 (4) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paget's disease of nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Lacunar stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device issue (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device loosening (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Methotrexate (N=216) | Period 1: Upadacitinib 15 mg (N=217) | Period 1: Upadacitinib 30 mg (N=215) | Periods 1+2: Upadacitinib 15 mg (N=318) | Periods 1+ 2: Upadacitinib 30 mg (N=311) | Period 2: Upadacitinib 15 mg Switched From Upadacitinib 30 mg (N=205)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 20 (27) | 18 (20) | 7 (7)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3) | 9 (17) | 18 (27) | 3 (4)
Bronchitis (Infections and infestations) | 7 (7) | 4 (4) | 4 (4) | 39 (50) | 40 (45) | 5 (5)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 21 (21) | 2 (2) | 20 (20)
Herpes zoster (Infections and infestations) | 1 (1) | 3 (3) | 5 (5) | 32 (33) | 32 (35) | 6 (6)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 15 (15) | 18 (19) | 2 (2)
Latent tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 25 (25) | 16 (16) | 5 (5)
Nasopharyngitis (Infections and infestations) | 7 (7) | 4 (4) | 4 (5) | 56 (79) | 38 (65) | 7 (8)
Upper respiratory tract infection (Infections and infestations) | 13 (16) | 9 (9) | 6 (6) | 38 (64) | 46 (66) | 5 (5)
Urinary tract infection (Infections and infestations) | 5 (5) | 10 (11) | 10 (12) | 43 (69) | 47 (87) | 13 (17)
Alanine aminotransferase increased (Investigations) | 3 (4) | 3 (3) | 5 (5) | 17 (27) | 23 (34) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 11 (15) | 19 (29) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 5 (5) | 9 (9) | 32 (57) | 58 (81) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 18 (19) | 20 (23) | 5 (5)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 10 (11) | 1 (1) | 5 (5) | 45 (60) | 29 (39) | 9 (11)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2) | 4 (4) | 8 (10) | 20 (24) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 5 (5) | 0 (0) | 28 (30) | 25 (26) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT02706951/Prot_002.pdf
  • Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT02706951/SAP_003.pdf